CLINICAL TRIAL: NCT01338285
Title: Studies of Myeloid Progenitor Cells in Workers Exposed to Formaldehyde, a Putative Leukemogen
Brief Title: Association of Formaldehyde Exposure to Myeloid Leukemia in Workers in Guangdong, China
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906178; 06-C-N178; NCT00516763 (obsolete NCT alias); NCT01338181 (obsolete NCT alias)
Record Dates: First submitted 2011-04-16; First posted 2011-04-19 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Epidemiology; Industrial Hygiene; Neoplasms
Keywords: Industry Hygiene; Molecular Epidemiology; Cancer Susceptability; Genotoxocity; FISH
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Workers exposed to high levels of formaldehyde and unexposed workers in Guangdong Province, China.

SUMMARY:
Background:

* Research suggests that occupational exposure to formaldehyde is associated with increased risk for myeloid leukemia, but the significance of these findings is uncertain because of inconsistencies among studies and lack of knowledge of how formaldehyde can cause leukemia.
* Damage to the DNA of myeloid cells (type of white blood cell) or an environmental factor not affecting the cell genetic machinery may be involved.

Objective: To determine if formaldehyde exposure is associated with genetic or other changes in myeloid cells.

Eligibility: Workers exposed to high levels of formaldehyde and unexposed workers in Guangdong Province, China.

Design:

* 40 exposed workers and 40 unexposed workers will be enrolled.
* Subjects wear small instruments at work that measure chemicals in the air for 1 or 2 days.
* Subjects have a brief physical examination and provide blood, urine, and mouth rinse samples.
* Subjects answer a questionnaire about work, smoking and drinking, use of medicines, medical history, general health, exposure to radiation and exposure to various substances at home.

DETAILED DESCRIPTION:
Research in industrial workers and professionals exposed to formaldehyde suggests that occupational exposure to this important chemical is associated with increased risk for myeloid leukemia. The significance, however, of these observations for occupational and environmental health is uncertain because of inconsistencies among epidemiologic studies and lack of a demonstrated mechanism through which formaldehyde can cause leukemia. Cytogenetic damage is one potential leukemogenic mechanism, but there are few studies of formaldehyde-exposed humans. Some experimental data suggest that epigenetic changes in myeloid cells could also be involved. We plan to study 40 workers exposed to high levels of formaldehyde and 40 unexposed controls to examine the hypothesis that formaldehyde is associated with these changes. To determine formaldehyde exposure, we will incorporate a number of methods, including questionnaires to determine potential past exposure and on-site monitoring to determine current average and peak intensities of exposure. We will then examine differences in aneuploidy and structural abnormalities in myeloid progenitor cells cultured from peripheral blood. We will specifically look for differences in genes associated with myeloid leukemia such as monosomy 7 and trisomy 8 using interphase and Octochrome FISH. We will also determine whether aberrant methylation in progenitor cells, specifically hypermethylation of genes associated with myeloid leukemia, is higher in those exposed to formaldehyde. This study will substantially contribute to our understanding of the leukemogenic potential of formaldehyde, which has important public health and regulatory implications.

ELIGIBILITY:
* Subjects will be recruited from a factory that manufactures plastic utensils and that has had a stable manufacturing process for the past five years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We identified one factory that produced formaldehyde-melamine resins and one factory that used formaldehyde-melamine resins to manufacture plastic utensils. Monitoring of formaldehyde levels was performed in these factories during an initial screening and it was established that there were no other exposures to known or suspected leukemogens or hematotoxicants (e.g., benzene, phenol, chlorinated solvents). We selected a control population from three workplaces in the same @@@geographic region as factories with formaldehyde exposure and enrolled workers who had comparable demographic and socioeconomic characteristics and who were engaged primarily in manufacturing. Detailed inspection of the control workplaces did not identify potential for occupational exposure to formaldehyde or any other@@@hematotoxic or genotoxic chemicals in excess of exposure levels in the general population.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2006-06-10 (Actual); Primary Completion 2007-05-01 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Hematotoxicity change | 2006-2034
  This study will determine if formaldehyde is associated with epigenetic changes in myeloid progenitor cells, including global methylation and hypermethylation in genes that have been linked to myeloid leukemia (ML) such as p15, HIC1, ER, CDH1 and ABL.
Leukemia-specific chromsome change | 28 years
  This study will determine if formaldehyde exposure is associated with aneuploidy in myeloid progenitor cells using interphase-FISH, with a particular focus on monosomy of chromosome 7 and aneuploidy of other relevant chromosomes, such as trisomy 8; and if formaldehyde exposure is associated with increased levels of structural aberrations relevant for myeloid leukemogenesis [e.g., 5q-] in myeloid progenitor cells using OctoChrome FISH, which will evaluate aberrations in all 24chromosomes.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Lan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Guangdong National Poison Control Center (NPCC), Guangzhou, China

REFERENCES:
- [Background] Cogliano VJ, Grosse Y, Baan RA, Straif K, Secretan MB, El Ghissassi F; Working Group for Volume 88. Meeting report: summary of IARC monographs on formaldehyde, 2-butoxyethanol, and 1-tert-butoxy-2-propanol. Environ Health Perspect. 2005 Sep;113(9):1205-8. doi: 10.1289/ehp.7542. PMID 16140628
- [Background] Hauptmann M, Lubin JH, Stewart PA, Hayes RB, Blair A. Mortality from lymphohematopoietic malignancies among workers in formaldehyde industries. J Natl Cancer Inst. 2003 Nov 5;95(21):1615-23. doi: 10.1093/jnci/djg083. PMID 14600094
- [Background] Egle JL Jr. Retention of inhaled formaldehyde, propionaldehyde, and acrolein in the dog. Arch Environ Health. 1972 Aug;25(2):119-24. doi: 10.1080/00039896.1972.10666147. No abstract available. PMID 5045063